CLINICAL TRIAL: NCT04623762
Title: Effect Of Yoga On Dyspnea, Sleep And Fatıgue In Chronıc Respıratory Dıseases
Brief Title: Yoga On Dyspnea, Sleep And Fatıgue In Chronıc Respıratory Dıseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, gülcan bahcecioğlu, ASSISTANT PROFESSOR, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020/4
Record Dates: First submitted 2020-10-29; First posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Chronic Respiratory Disease
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): yoga was not done
- Experimental group (Experimental): yoga was done
  Interventions: Other: Yoga

INTERVENTIONS:
Other: Yoga — yoga application
  Arms: Experimental group

SUMMARY:
Although there are a limited number of studies in the literature investigating the effect of yoga on dyspnea, quality of life and respiratory functions of chronic respiratory patients There is no study examining the effect of yoga on sleep and fatigue of chronic respiratory patients. Therefore, this study was conducted to determine the effect of yoga on dyspnea, sleep, and fatigue applied to chronic respiratory patients.

DETAILED DESCRIPTION:
Chronic respiratory diseases (CSFD) are chronic diseases of the airways and other structures of the lung. Two of the most common of these diseases are asthma and chronic obstructive pulmonary disease. Asthma and chronic obstructive pulmonary disease (COPD); mortality, morbidity and prevalence of chronic respiratory diseases are increasingly increasing across countries. COPD; It has been defined as a common, preventable and treatable disease characterized by permanent airflow restriction, which is associated with the increased chronic inflammatory response of the airways and lungs to harmful gases and particles Every year, 3 million people die of COPD in the world and this rate constitutes 6% of all deaths If it is asthma; It is defined as a heterogeneous disease characterized by chronic airway inflammation associated with airway hyperresponsiveness to direct or indirect stimuli. Asthma is seen at a rate of 1-18% in the whole world population

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-55 and diagnosed with asthma and COPD for at least six months,

  * Do not have any disease that causes insomnia and do not use sleeping pills
  * Has the ability to use the internet actively, download the ZOOM program to the phone or computer and participate in the application.

Have not participated in a similar regular exercise program in the last 6 months,

* Do not have any respiratory system disease other than asthma and COPDY,
* Not in exacerbation period,
* Do not have a physical illness or cognitive deficiency and a psychiatric disease that prevents understanding of the education given,
* Patients who were literate and volunteered to participate in the study were included in the study.

Exclusion Criteria:

* In the period of exacerbation Have participated in a similar regular exercise program in the last 6 months, Those who cannot download the ZOOM program and participate in the application

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-07-28 (Actual)

PRIMARY OUTCOMES:
Chronic Obstructive Pulmonary Disease and Asthma Fatigue Scale | Change from Baseline Fatigue at 2 months
  Revicki et al. (2010) to determine the effect of COPD and asthma on fatigue. Cronbach's alpha value of the scale was found to be 0.95. The scale, which consists of 12 items, is a five-point Likert type, and the minimum total score that can be obtained from the scale is 12 and the maximum total score is 60. The higher the score obtained from the scale indicates that the fatigue level of the person is high. Turkey on the scale of the Turkish validity and reliability study of Arslan and by Öztunç (2013) was determined to be conducted and Cronbach's alpha values for the reliability coefficient of 0.92.

SECONDARY OUTCOMES:
Asthma and COPD Sleep Scale (CASIS) | Change from Baseline Sleep at 2 months
  It was developed by Pokrzywinski et al. (2009) to reveal the effect of asthma and COPD disease on sleep. The Cronbach Alpha Coefficient of the scale was found to be 0.90. The Turkish validity and reliability study of the scale was conducted by Ayhan and Kıyak (2011) and the cronbach alpha coefficient was determined as 0.87. The items of the questions in the scale consisting of 7 questions in total are likert in the form of never, rarely, sometimes, often, and very often.

OTHER OUTCOMES:
Medical Research Board Dyspnea Scale (MRC): | Change from Baseline MRC at 2 months
  t is a five-item scale developed by the British Medical Research Board for the evaluation of dyspnea. While applying the Medical Research Council Dyspnea Scale, patients are asked to indicate the activity level that causes dyspnea. The patient chooses the most appropriate level that defines the respiratory distress by reading the options on the scale. The options are graded from 0 to 4; 0 points, no dyspnea; 1 point of mild dyspnea (respiratory distress when moving fast on a flat surface and climbing slightly uphill); 2 points of moderate dyspnea (walk slower than peers when walking on a flat surface, pausing to breathe); 3 points are scored as severe dyspnea (stopping to breathe after walking for 100 meters or a few minutes) and 4 points as very severe dyspnea (breathlessness while wearing clothes, taking off or going to the toilet while doing daily work at home).
Pulmonary Functions Monitoring Form | Change from Baseline Pulmonary Functions at 2 months
  Pulmonary function tests are evaluated with the spirometer to determine the degree of airway limitation and whether it is reversible and to diagnose asthma. Forced vital capacity (FVC), forced expiratory volume in one second (FEV1), highest expiratory flow rate (PEF) and FEV1 / FVC measurements were evaluated to evaluate its restriction.

CONTACTS AND LOCATIONS:
Overall Officials: Gülcan Bahçecioğlu Turan, Principal Investigator — Fırat Universty
Locations (2):
- Turkey (Türkiye) (2):
  - Fırat university, Erzurum, Center
  - Sabahattin Zaim University, Istanbul, Center

IPD SHARING:
Plan to Share IPD: No